CLINICAL TRIAL: NCT01547585
Title: A Randomized Controlled Trial to Determine the Low Density Lipoprotein Cholesterol (LDL-C) Lowering Effect of Whole Soy: a Dose Response Study
Brief Title: A Human Trial to Assess the Low Density Lipoprotein Cholesterol (LDL-C) Lowering Effect of Soy
Acronym: SOY-LDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guelph Food Research Centre (Other Government)
Collaborators: University of Guelph (Other); Glycemic Index Laboratories, Inc (Industry); Canadian Centre for Agri-Food Research in Health and Medicine (Other)
Responsible Party: Principal Investigator, Dan Ramdath, Principal Investigator, Guelph Food Research Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SOY-CVD-2012; RBPI#1746 (Other Grant/Funding Number: Adriculture and Agri-Food Canada)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hypercholesterolemia; Cardiovascular Disease; CRP
Keywords: Cholesterol; Cardiovascular disease; Soy; Dose-response
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): - Isocaloric control muffins
  Interventions: Other: Standardized soy containing muffin
- Low Dose Soy (Experimental): - Isocaloric muffins containing low dose of soy
  Interventions: Other: Standardized soy containing muffin
- High Dose Soy (Experimental): - Isocaloric muffins containing high dose soy
  Interventions: Other: Standardized soy containing muffin

INTERVENTIONS:
Other: Standardized soy containing muffin — Standardized muffin containing two levels of soy
  Other Names: Soy containing muffins

SUMMARY:
This study is being conducted to test the hypothesis that daily consumption of a baked food product containing whole soy for 6 weeks will significantly reduce plasma Low Density Lipoprotein Cholesterol (LDL-C) in individuals with hypercholesterolemia. As such the overall goals of this study are to determine whether daily consumption of muffins made from whole soy flour for 6 weeks can lower plasma LDL-Cholesterol, and if so, establish whether the effect is dose-dependent. To do this, study collaborators will: (1) conduct a detailed chemical and physical characterization of certified defatted whole soy flour that will be incorporated into a muffin; (2) formulate and produce a palatable whole soy flour muffin along with a control muffin containing wheat flour; (3) conduct a parallel controlled trial in which soy muffins will be fed randomly to persons with elevated LDL-cholesterol in a human clinical trial. All participants will be randomized into one of three groups and asked to eat two muffins daily for 6 weeks in the following combination: high dose soy; control group or low dose soy. Before, after, and mid-way during the feeding period, blood samples will be obtained for measurements of lipids, glucose, insulin, inflammation, and soy phytochemicals. The effect of soy consumption on waist circumference, body mass index (BMI) and blood pressure will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (not pregnant or lactating) aged 30-70 year
* Body mass index (BMI) ≤40kg/m² and ≥18.5kg/m²
* Fasting plasma total cholesterol ≥5.0
* Fasting plasma LDL cholesterol ≥3.0 and <5.0 mmol/L.

Exclusion Criteria:

* Fasting plasma triglycerides ≥4.0 mmol/L
* Abnormal liver and kidney function
* Unstable body weight(>3kg change in 3 months) or intention to lose or gain weight;
* Diabetes mellitus (fasting plasma glucose ≥7.0 mmol/L or use of insulin or any hypoglycemic or anti-hyperglycemic medication);
* Use of any prescription or non-prescription drug, prebiotics or probiotics, herbal or nutritional supplement known to affect blood lipids, except for stable doses (no change in 3 months) of thyroxine, oral contraceptive agents, hormone replacement therapy, and medications for controlling blood pressure);
* Major surgical or medical events within the past 3 months;
* Presence of a gastrointestinal disorder or medication that alters the digestion and absorption of nutrients; including antibiotic use within the past 6 weeks.
* Consumption of a diet containing ≥15% of energy from saturated fat;
* Any food allergy or aversion or unwillingness to eat wheat, soy or milk;
* Consumption of ≥5 servings per week of soy based food products;
* Consumption of an average of >2 alcoholic beverages per day;
* Regular smokers (smoking ≥1 cigarette per day) of cigarettes or cigars

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein Cholesterol (LDL-Cholesterol) | 6 weeks

SECONDARY OUTCOMES:
high sensitivity c-reactive protein (hsCRP) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alison Duncan, PhD, RD, Principal Investigator — University of Guelph; Thomas Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc; Heather Blewett, PhD, Principal Investigator — Canadian Centre for Agri-Food Research in Health and Medicine
Locations (3):
- Canada (3):
  - Canadian Centre for Agri-food Research in Health and Medicine, Winnipeg, Manitoba
  - Human Nutraceutical Research Unit. University of Guelph, Guelph, Ontario
  - Glycemic Index Laboratories, Inc, Toronto, Ontario

REFERENCES:
- [Background] Reinwald S, Akabas SR, Weaver CM. Whole versus the piecemeal approach to evaluating soy. J Nutr. 2010 Dec;140(12):2335S-2343S. doi: 10.3945/jn.110.124925. Epub 2010 Oct 27. PMID 20980652
- [Background] Zhang X, Shu XO, Gao YT, Yang G, Li Q, Li H, Jin F, Zheng W. Soy food consumption is associated with lower risk of coronary heart disease in Chinese women. J Nutr. 2003 Sep;133(9):2874-8. doi: 10.1093/jn/133.9.2874. PMID 12949380
- [Background] Kokubo Y, Iso H, Ishihara J, Okada K, Inoue M, Tsugane S; JPHC Study Group. Association of dietary intake of soy, beans, and isoflavones with risk of cerebral and myocardial infarctions in Japanese populations: the Japan Public Health Center-based (JPHC) study cohort I. Circulation. 2007 Nov 27;116(22):2553-62. doi: 10.1161/CIRCULATIONAHA.106.683755. Epub 2007 Nov 19. PMID 18025534
- [Background] Nanri A, Mizoue T, Takahashi Y, Kirii K, Inoue M, Noda M, Tsugane S. Soy product and isoflavone intakes are associated with a lower risk of type 2 diabetes in overweight Japanese women. J Nutr. 2010 Mar;140(3):580-6. doi: 10.3945/jn.109.116020. Epub 2010 Jan 6. PMID 20053935
- [Background] Yang B, Chen Y, Xu T, Yu Y, Huang T, Hu X, Li D. Systematic review and meta-analysis of soy products consumption in patients with type 2 diabetes mellitus. Asia Pac J Clin Nutr. 2011;20(4):593-602. PMID 22094845
- [Background] Anderson JW, Bush HM. Soy protein effects on serum lipoproteins: a quality assessment and meta-analysis of randomized, controlled studies. J Am Coll Nutr. 2011 Apr;30(2):79-91. doi: 10.1080/07315724.2011.10719947. PMID 21730216
- [Background] Anderson JW, Johnstone BM, Cook-Newell ME. Meta-analysis of the effects of soy protein intake on serum lipids. N Engl J Med. 1995 Aug 3;333(5):276-82. doi: 10.1056/NEJM199508033330502. PMID 7596371
- [Background] Zhan S, Ho SC. Meta-analysis of the effects of soy protein containing isoflavones on the lipid profile. Am J Clin Nutr. 2005 Feb;81(2):397-408. doi: 10.1093/ajcn.81.2.397. PMID 15699227
- [Background] Dewell A, Hollenbeck PL, Hollenbeck CB. Clinical review: a critical evaluation of the role of soy protein and isoflavone supplementation in the control of plasma cholesterol concentrations. J Clin Endocrinol Metab. 2006 Mar;91(3):772-80. doi: 10.1210/jc.2004-2350. Epub 2005 Dec 29. PMID 16384855
- [Background] Sirtori CR, Eberini I, Arnoldi A. Hypocholesterolaemic effects of soya proteins: results of recent studies are predictable from the anderson meta-analysis data. Br J Nutr. 2007 May;97(5):816-22. doi: 10.1017/S0007114507670810. PMID 17408521
- [Background] Sacks FM, Lichtenstein A, Van Horn L, Harris W, Kris-Etherton P, Winston M; American Heart Association Nutrition Committee. Soy protein, isoflavones, and cardiovascular health: an American Heart Association Science Advisory for professionals from the Nutrition Committee. Circulation. 2006 Feb 21;113(7):1034-44. doi: 10.1161/CIRCULATIONAHA.106.171052. Epub 2006 Jan 17. PMID 16418439
- [Background] Klein MA, Nahin RL, Messina MJ, Rader JI, Thompson LU, Badger TM, Dwyer JT, Kim YS, Pontzer CH, Starke-Reed PE, Weaver CM. Guidance from an NIH workshop on designing, implementing, and reporting clinical studies of soy interventions. J Nutr. 2010 Jun;140(6):1192S-1204S. doi: 10.3945/jn.110.121830. Epub 2010 Apr 14. PMID 20392880
- [Derived] Padhi EM, Blewett HJ, Duncan AM, Guzman RP, Hawke A, Seetharaman K, Tsao R, Wolever TM, Ramdath DD. Whole Soy Flour Incorporated into a Muffin and Consumed at 2 Doses of Soy Protein Does Not Lower LDL Cholesterol in a Randomized, Double-Blind Controlled Trial of Hypercholesterolemic Adults. J Nutr. 2015 Dec;145(12):2665-74. doi: 10.3945/jn.115.219873. Epub 2015 Oct 7. PMID 26446482